CLINICAL TRIAL: NCT02692118
Title: Inflammatory Mediators in Sepsis as Indicator for Infection vs Inflammation
Brief Title: Inflammatory Mediators in Early Sepsis
Acronym: Tusep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: AnaTubingen
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sepsis: Patients with septic shock admitted to ICU

SUMMARY:
Sepsis is still a challenge for clinicians since the detailed pathomechanism are still unknown and until now early markers for sepsis are not defined yet. Immunological pathways and new mediators defined in animal models are not yet investigated in patients with sepsis. Therefore the investigators will measure new mediators in patients with septic shock.

DETAILED DESCRIPTION:
Semaphorins 1 to 7 will be determined in Blood of patients with early septic shock. Concentration will be compared with blood concentration of postoperative patients suffering systemic inflammatory response syndrome (SIRS).

ELIGIBILITY:
Inclusion Criteria:

* Septic Shock

Exclusion Criteria:

* Age < 18 > 85
* no consent of caregiver
* Trauma patients
* Burn patients
* Immunosuppression
* Pregnancy
* HIV- hepatitis infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care patients with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Semaphorin 1 to 7 in plasma of septic patients | 12 months
  Concentration of Semaphorin in plasma of 60 sepsis patients [pg/ml].

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Granja T, Kohler D, Tang L, Burkard P, Eggstein C, Hemmen K, Heinze KG, Heck-Swain KL, Koeppen M, Gunther S, Blaha M, Magunia H, Bamberg M, Konrad F, Ngamsri KC, Fuhr A, Keller M, Bernard AM, Haeberle HA, Bakchoul T, Zarbock A, Nieswandt B, Rosenberger P. Semaphorin 7A coordinates neutrophil response during pulmonary inflammation and sepsis. Blood Adv. 2024 Jun 11;8(11):2660-2674. doi: 10.1182/bloodadvances.2023011778. PMID 38489236